# The Ohio State University Consent to Participate in Research

Study Title: Survivorship ECHO Project with Ohio State University

**Comprehensive Cancer Center- James Cancer Hospital** (OSUCCC-James) and Ohio State University Network

Protocol Number: 2021C0115

Researcher: Ashley Pariser, MD

**Sponsor:** The Ohio State University

This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate.

# Your participation is voluntary.

Please consider the information carefully. Feel free to ask questions before making your decision whether or not to participate.

### **Purpose:**

The purpose of the Survivorship ECHO Project is to deliver education and support to healthcare providers regarding best practices in cancer survivorship to assist in caring for cancer patients. The education is provided in the Project ECHO format which will be on Zoom.

#### Procedures/Tasks:

You are eligible to participate in this research if you are age 18 or older. You must be a healthcare worker in the field of cancer. People taking part in the project will be asked to attend 6 hour-long Zoom conference-based lectures with case-based discussion. Participants will be asked to complete two online surveys prior to the first educational session, and two post-curriculum surveys (one at the conclusion of the curriculum, and one approximately six months later.

We will collect and confirm contact information such as email address to ensure participants receive the online surveys. Each survey should take about 10 minutes to complete. We will ask questions about participant knowledge of cancer survivorship as well as self-efficacy, or confidence in your ability to address cancer survivors' concerns. You do not have to finish the project surveys in one sitting. You are able to go back into the surveys at a later time and pick up where you left off. You are free to skip any question you do not want to answer. Just select "prefer not to answer" on the surveys.

This project will also ask your institution to provide aggregate-level data from the electronic medical record system to evaluate changes in clinical care of breast cancer survivors before and after this educational component implementation. The privacy of breast cancer patients and the participants of this study (the providers) will be protected at all times; OSU will receive de-identified, summary data only with no link to identifying information. Evaluation measures will look at screening rates among the clinical care of breast cancer survivors, as well as rates of referrals to specialists and communications between oncology providers and primary care. At the conclusion of the project, a summary of the evaluation will be provided to participants via the email provided for participation.

#### **Duration:**

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

#### **Risks and Benefits:**

You may benefit directly from this study by increasing your knowledge and self-efficacy in caring for cancer survivors.

There are no physical risks, pain or discomfort involved in taking part in the project. This is a research study that is providing education and asking questions to assess perceived knowledge and self-efficacy levels. However, if you are bothered by a question, you have the right to not answer the question or select "prefer not to answer." You can stop taking part in the project at any time.

# Confidentiality:

We will work to make sure that no one sees your online responses without approval. But, because we are using the Internet, there is a chance that someone could access your online responses without permission. In some cases, this information could be used to identify you. Your data will be protected with a code to reduce the risk that other people can view the responses.

Also, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law. Also, your records may be reviewed by the following groups (as applicable to the research):

- Office for Human Research Protections or other federal, state, or international regulatory agencies;
- The Ohio State University Institutional Review Board or Office of Responsible Research Practices;

- Authorized Ohio State University staff not involved in the study may be aware that you are participating in a research study and have access to your information; and
- The sponsor, if any, or agency (including the Food and Drug Administration for FDA-regulated research) supporting the study.

#### **Future Research:**

Your de-identified information will not be used or shared for future research.

### **Incentives:**

Participants will receive a \$25 gift card after completing the baseline survey and a \$25 gift card after completing the end-of-curriculum survey. Gift cards are distributed via email to the email address used for study participation. By law, payments to participants are considered taxable income.

### **Participant Rights:**

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By agreeing to participate, you do not give up any personal legal rights you may have as a participant in this study.

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of participants in research.

### **Contacts and Ouestions:**

For questions, concerns, or complaints about the study, or you feel you have been harmed as a result of study participation, you may contact Ashley Pariser, MD at 614-366-8541 or Ashley.Pariser@osumc.edu.

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251 or hsconcerns@osu.edu.

## **Providing consent**

I have read (or someone has read to me) this page and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study. I am not giving up any legal rights by agreeing to participate.

To print or save a copy of this page, select the print button on your web browser.

Please click the button below to proceed and participate in this study. If you do not wish to participate, please close out your browser window.